CLINICAL TRIAL: NCT01907984
Title: Preoperatively Administered Single Dose Diclofenac Reduces the Intensity of Acute Postcraniotomy Headache and Decreases Postoperative Analgesic Requirements- a Randomized, Controlled Trial
Brief Title: Diclofenac Administered Before Skull Operations Reduces the Severity of Headache After the Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, assistant lecturer anesthesiologist and intensive care specialist, University of Debrecen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5481-1/2013/EKU; DEOEC RKEB/IKEB:3769-2012 (Other: University of Debrecen,RKEB/IKEB)
Record Dates: First submitted 2013-07-11; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Postcraniotomy Headache; Intraoperative Analgesic Use; Postoperative Analgesic Use; Postoperative Complications
Keywords: premedication; diclofenac; postoperative headache; Visual Analog Scale
MeSH Terms: conditions — Postoperative Complications | interventions — Diclofenac; Midazolam

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac and Midazolam (Experimental): Diclofenac 100 mg tablet and Midazolam 7.5 mg tablet were administered by mouth as premedication 30 minutes before surgical interventions.
  Interventions: Drug: Diclofenac; Drug: Midazolam
- Midazolam (Active Comparator): Midazolam 7.5 g tablet was administered as premedication by mouth 30 minutes before surgical interventions.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Diclofenac
  Other Names: DICLOFENAC-ratiopharm; Voltaren; DICLOFENAC-STADA
  Arms: Diclofenac and Midazolam
Drug: Midazolam
  Other Names: Dormicum

SUMMARY:
Purpose:

According to the proposal of the International Headache Society acute postcraniotomy headache (PCH) is defined as a headache of variable intensity, being most serious at the site of surgical intervention and developing within 7 days after craniotomy. Typically, pain resolves within 3 months after surgery. According to the literature the incidence of acute PCH during the postoperative period is 60% among patients undergoing elective craniotomies. No standardized international guidelines are available on the treatment of PCH to the present day. Treatment methods can be different based on the country and institution where they are used, or even physicians individually can have distinct medication regime, which sometimes happens to be habitual and lacks clinical evidences.

The Department of Anesthesiology and Intensive Care Medicine at the University of Debrecen has been giving 100 mg diclofenac with analgesic purpose, as part of the premedication to neurosurgical patients for several years. It was observed that the postoperative headache following craniotomy was milder comparing to data published in the international literature. A pilot study was carried out with similar settings which found the that incidence of PCH was lower and less analgesics were required without any further unwanted side-effects among patients who received 100 mg diclofenac as part of the premedication.

Hypothesis:

100 mg preoperatively given diclofenac significantly reduces the incidence and severity of postcraniotomy headache.

DETAILED DESCRIPTION:
Before surgery, every patient's previous history was taken routinely and along with this, special attention was paid to a history of preoperative headache, its severity and any analgesics used regularly prior to surgery. In this study 200 cooperative adults (over 18 years) undergoing elective craniotomy were randomly assigned into two groups with: 100 patients received 7.5 mg midazolam and 100 mg diclofenac as premedication, while the other 100 members of the control group received only 7.5 mg midazolam one hour prior to surgery. Envelop randomization was used to schedule patients to diclofenac or to placebo groups. Neither the anesthetists, nor the physician obtaining the postoperative VAS scores were aware of the actual patient's grouping (diclofenac or placebo) during the entire study. For induction of anesthesia, we used propofol (1-2,5 mg/kgBW), whereas for maintenance of anesthesia we used the combination of fentanyl, rocuronium, and sevoflurane. Craniotomy and opening the dura occurred always after the tissue saturation of sevoflurane and low-flow anesthetic technique was applied at a sevoflurane concentration ranging from 1.2 to 2.1 V% as required for maintenance of adequate anesthesia. Fentanyl was administered as an initial bolus of 100-150 µg followed by a maintenance dose of 2 µg/kgBW/h. The total dose of fentanyl was calculated offline after the procedure in all cases. The surgical site was infiltrated by a combination of 2% lidocaine and epinephrine in all cases. All patients were admitted to the neurosurgical ICU for postoperative observation. A stepwise analgesic regimen was decided prior the study. Severity of pain was assessed regularly by the ICU nurses and additional analgesics were used if the patient complained a headache severity of VAS >3. In these cases additional paracetamol (1-2 g given intravenously) was administered. If this was not effective, an additional dose of 100 mg diclofenac was given to the patients. In case of further ineffectivity, tramadol was administered in a dose of 100 mg per os or iv. At the end of the study the cumulative dose of analgesics that was administered to the patients was calculated. For sake of clarity we transformed analgesic doses to equianalgetic doses of intramuscular morphine according to the table of the Oxford Pain Site and these values were used for further comparisons of analgesic requirements.

Pain assessment occurred at bedrest state by using a 0-10 scaled visual analogue scale (VAS). Assessment of actual VAS scores was regularly performed by the nurses of the neurosurgical ICU during days 1-5 and rescue analgesics were given according to the actual needs of the patients. An independent physician (who was unaware of randomization) performed an additional check of VAS scores by asking the patient, what was her/his worse pain during the day. As the patient's satisfaction was considered to be dependent on the worse pain, only these VAS scores were used for further analysis.

The investigators intended to answer the following study questions:

* Our research intended to examine whether 100 mg preoperatively give diclofenac reduces the incidence and severity of PCH on the first and fifth postoperative days.
* Is there a difference in the incidence and severity of PCH between patients who underwent infra- or supratentorial interventions?
* Does 100 mg preoperatively give diclofenac reduce intraoperative and postoperative analgesic needs?
* Does 100 mg preoperatively give diclofenac increase the incidence of postoperative hemorrhagic events?

Grouping of the patients:

The anesthesiologist on duty assigned the participants randomly to the control or to the diclofenac group by using envelope randomization technique the day before the surgery.

Members of the control group received 7.5 mg midazolam, while members of the diclofenac group received 7.5 mg midazolam and 100 mg diclofenac for premedication.

Gathering data:

Since no objective method exist to measure pain patients were asked to rate their headache subjectively with the help of a visual analog scale, where 0 stands for no pain and 10 for intolerable pain. In order to make the interpretation of data easier the scale was divided into three parts: between 1 and 3 the headache is mild, from 4 to 6 it is moderate, while 7 or a greater value represents a particularly strong pain.

The sites of the surgical intervention, intra- and postoperative analgesic needs, postoperative complications were recorded individually onto a personal data sheet.

Each data mentioned above was registered by a third pre-trained, independent (blind) member of the study team, who was unaware of the premedication and grouping of patients.

Statistical methods:

Statistical analysis was performed using Statistica for Windows (Statsoft, Tulsa, USA) statistical program. A normality test revealed that data of VAS scores and analgesic requirements show non-normal distribution, therefore a non-parametric Mann-Whitney test was used for further comparisons. A p-value of <0.05 was accepted as statistically significant during analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were over the age of 18, able to cooperate and underwent elective craniotomy at the Department of Neurosurgery of the University of Debrecen.
* Patients with full awareness and without existing sensory or severe motor aphasia at admission or postoperatively.
* After written informed consent and written agreement was obtained from each participant.

Exclusion Criteria:

* Patients under the age of 18, patients who were unable to cooperate and who underwent traumatic or emergency interventions.
* Patients taking non-steroidal anti-inflammatory agents prior to surgery for any reasons were excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Severity of headache was measured with Visual Analog Scale (VAS) | Changes from Baseline in Visual Analog Scale assessed at the first postoperative day
  Severity of pain was assessed using a visual analogue scale 24 hours preoperatively, on the day of surgery 30 minutes before the operation, the current severity of headache on the first and fifth postoperative days and the strongest pain experienced since the last Visual Analog Scale assessments.
Severity of headache was measured with Visual Analog Scale (VAS) | Changes from Baseline in Visual Analog Scale assessed at the 5. postoperative day
  Severity of pain was assessed using a visual analogue scale 24 hours preoperatively, on the day of surgery 30 minutes before the operation, the current severity of headache on the first and fifth postoperative days and the strongest pain experienced since the last Visual Analog Scale assessments.

SECONDARY OUTCOMES:
Severity of postcraniotomy headache within supra- and infratentorial sub-groups. | Changes from Baseline in Visual Analog Scale assessed at the first and fifth postoperative day
  Patients were sub-grouped according to the site of the surgical intervention, either supra- or infratentorial skull surgery, the severity of PCH was measured among these groups by means of Visual Analog Scale.

OTHER OUTCOMES:
Analgesic need during the first five postoperative days. | Participants were followed for 5 days postoperatively
  The total amount of analgesics administered were recorded during the first five postoperative days and then converted into intramuscular morphine equivalents.
Postoperative complications during the first five postoperative days | Participants were followed for 5 days postoperatively
  Postoperative complications such as bleeding at the surgical site, gastrointestinal problems or kidney dysfunctions were also registered.
Intraoperative fentanyl use | Participants were followed during the operation on day 1.
  Intraoperative fentanyl use was registered as micrograms per kilogram body weight and micrograms per hour as well.

CONTACTS AND LOCATIONS:
Overall Officials: Csilla Molnár, MD, PhD, Principal Investigator — University of Debrecen Medical and Health Science Center Department of Anesthesiology and Intensive Care 4032-Debrecen, Nagyerdei krt 98. Hungary Tel/fax: +36-52-255-347
Locations (1):
- University of Debrecen Medical and Health Science Center Department of Anesthesiology and Intensive Care, Debrecen, Hajdú-Bihar, Hungary

REFERENCES:
- [Background] De Benedittis G, Lorenzetti A, Migliore M, Spagnoli D, Tiberio F, Villani RM. Postoperative pain in neurosurgery: a pilot study in brain surgery. Neurosurgery. 1996 Mar;38(3):466-9; discussion 469-70. doi: 10.1097/00006123-199603000-00008. PMID 8837797
- [Background] Rocha-Filho PA, Gherpelli JL, de Siqueira JT, Rabello GD. Post-craniotomy headache: characteristics, behaviour and effect on quality of life in patients operated for treatment of supratentorial intracranial aneurysms. Cephalalgia. 2008 Jan;28(1):41-8. doi: 10.1111/j.1468-2982.2007.01465.x. Epub 2007 Nov 6. PMID 17986272
- [Background] Quiney N, Cooper R, Stoneham M, Walters F. Pain after craniotomy. A time for reappraisal? Br J Neurosurg. 1996 Jun;10(3):295-9. doi: 10.1080/02688699650040179. PMID 8799542
- [Background] Thibault M, Girard F, Moumdjian R, Chouinard P, Boudreault D, Ruel M. Craniotomy site influences postoperative pain following neurosurgical procedures: a retrospective study. Can J Anaesth. 2007 Jul;54(7):544-8. doi: 10.1007/BF03022318. PMID 17602040
- [Background] Nguyen A, Girard F, Boudreault D, Fugere F, Ruel M, Moumdjian R, Bouthilier A, Caron JL, Bojanowski MW, Girard DC. Scalp nerve blocks decrease the severity of pain after craniotomy. Anesth Analg. 2001 Nov;93(5):1272-6. doi: 10.1097/00000539-200111000-00048. PMID 11682413
- [Background] Gottschalk A, Berkow LC, Stevens RD, Mirski M, Thompson RE, White ED, Weingart JD, Long DM, Yaster M. Prospective evaluation of pain and analgesic use following major elective intracranial surgery. J Neurosurg. 2007 Feb;106(2):210-6. doi: 10.3171/jns.2007.106.2.210. PMID 17410701
- [Background] Gottschalk A, Yaster M. The perioperative management of pain from intracranial surgery. Neurocrit Care. 2009;10(3):387-402. doi: 10.1007/s12028-008-9150-3. Epub 2008 Oct 1. PMID 18830699
- [Background] Roberts GC. Post-craniotomy analgesia: current practices in British neurosurgical centres--a survey of post-craniotomy analgesic practices. Eur J Anaesthesiol. 2005 May;22(5):328-32. doi: 10.1017/s0265021505000554. PMID 15918378
- [Background] de Gray LC, Matta BF. Acute and chronic pain following craniotomy: a review. Anaesthesia. 2005 Jul;60(7):693-704. doi: 10.1111/j.1365-2044.2005.03997.x. PMID 15960721
- [Background] Umamaheswara Rao GS, Gelb AW. To use or not to use: the dilemma of NSAIDs and craniotomy. Eur J Anaesthesiol. 2009 Aug;26(8):625-6. doi: 10.1097/EJA.0b013e32832a21ad. No abstract available. PMID 19584610
- [Background] Schug SA, Manopas A. Update on the role of non-opioids for postoperative pain treatment. Best Pract Res Clin Anaesthesiol. 2007 Mar;21(1):15-30. doi: 10.1016/j.bpa.2006.12.002. PMID 17489217